CLINICAL TRIAL: NCT00665314
Title: A Multicenter, Randomized, Comparative, Patient-blinded Study to Evaluate the Safety and Efficacy of G-CSF Alone Versus AMD3100 (240 µg/kg) Added to a G-CSF Mobilization Regimen in Adult Patients With Non-Hodgkin's Lymphoma (NHL), Hodgkins Disease (HD) or Multiple Myeloma (MM) Who Have Previously Failed Stem Cell Collections or Collection Attempts
Brief Title: Evaluation of the Safety and Efficacy of the Addition of AMD3100 to a G-CSF Mobilization Regimen in Patients With Lymphoma (NHL and HD) and Multiple Myeloma (MM).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMD3100-EU23; EudraCT number: 2006-00424729
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Lymphoma; Non Hodgkin's Lymphoma; Hodgkin's Disease; Multiple Myeloma
Keywords: Mobilisation stem cells; G-CSF Mobilisation Regimen; Lymphoma; Multiple Myeloma; Adult patients with lymphoma (Non Hodgkin's Lymphoma, Hodgkin's Disease) or Multiple Myeloma who previously failed Stem Cell Collections or Collection attempts.
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma | interventions — plerixafor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMD3100 added to a G-CSF Mobilisation regimen (Experimental): AMD3100 added to a G-CSF Mobilisation regimen
  Interventions: Drug: Plerixafor (AMD3100)
- G-CSF plus placebo (Active Comparator): G-CSF plus placebo
  Interventions: Drug: Can be any registered nonpegylated form of G-CSF

INTERVENTIONS:
Drug: Plerixafor (AMD3100) — 0.24mg/kg SC for 2 to 7 days.
  Arms: AMD3100 added to a G-CSF Mobilisation regimen
Drug: Can be any registered nonpegylated form of G-CSF — 10mcg/kg SC for 4 days followed by an additional 2 to 7 days.
  Arms: G-CSF plus placebo

SUMMARY:
Some patients with multiple myeloma or lymphoma will need treatment with high dose chemotherapy to treat their condition. This potent treatment will kill many of the blood-forming cells in the bone marrow. The patient will therefore need these blood-forming cells replaced after the chemotherapy treatment. This is done by collecting some of teh patients own blood-forming stem cells before chemotherapy, storing them and then infusing them into the patient after chemotherapy (in the same way as a blood transfusion is given). The stem cells will then make their way unto the bone marrow and re-populate it. Having stem cells collected and returned later is called an "Autologous Transplant".

In most patients these blood-forming stem cells (which normally live in the bone marrow) are "mobilized" into the blood stream where they are then collected by a process called apheresis (a bit like donating blood). This process of mobilization is not always successful. In this study patients who did not collect enough stem cells in a previous cell collection attempt to have an autologous stem cell transplant will participate. Patients will be mobilized with G-CSF (current standard treatment to mobilize stem cells) and the effect of adding AMD3100 to G-CSF will be studied by comparing outcomes in patients who get G-CDF with placebo (non-active substance which looks like AMD3100) to patients who get G-CSF with AMD3100.

AMD3100 is a member of a new class of medications called "chemokine inhibitors". The drug triggers the movement of stem cells out of the bone marrow into the blood stream. In previous studies with healthy volunteers and cancer patients, when AMD3100 and G-CSF were used in combination, a greater number of stem cells were mobilized into the blood stream than by using g-CSF alone.

The purposes of this study are to measure how many stem cells can be collected, the number of days to collect those cells and the safety of a mobilization regimen of AMD3100 with G-CSF compared to G-CSF with placebo. If enough cells are collected to have a transplant, the study will also evaluate how well the cells grow when transplanted.

DETAILED DESCRIPTION:
This is a multicenter, randomized, comparative, patient-blinded study. Patients with NHL, HD or MM who would benefit from an autologous stem cell transplant, who failed previous collections or collection attempts with a mobilization regimen of chemotherapy with or wihoutG-CSF, and who meet the inclusion/exclusion criteria are eligible to receive AMD3100(240µg/kg) or placebo (both given as an evening dose).

Patients will undergo mobilization with G-CSF (10µg/kg) for 4 consecutive days. On Day 4, AMD3100 (240µg/kg) or placebo will be administered in the evening prior to the first apheresis and each subsequent evening prior to apheresis thereafter, such that there is a 10 to 11 hour interval between dosing and the initiation of apheresis. Patients will continue to receive G-CSF on each day of apheresis. G-CSF will be administered in the morning and approximately 1 hour prior to apheresis. Patients will undergo a minimum of 2 and a maximum of 7 aphereses until a minimum of 2x10^6 CD34+ cells/kg or greater than or equal to 5x10^6 CD34+cells/kg are collected. More cells may be collected, if done within the 7 aphereses. Patients who are to receive a tandem transplant will undergo a minimum of 2 and maximum of 7 aphereses until a minimum of 4x10^6 CD34+ cells/kg are collected. Aphereses should be performed on consecutive days (including weekend days)

The patient will have a peripheral blood (PB) sample collected to measure the number of CD34+ cell in PB at baseline prior to administration of G-CSF, prior to each administration of AMD3100 or placebo and at the initiation of apheresis. In addition, a sample will be obtained from each apheresis product to measure the number of CD34+ cells collected in the apheresis product.

Patients who fail to collect greater than or equal to 0.8x10^6 CD34+ cells/kg in 7 aphereses will be offered a rescue arm giving AMD3100 plus G-CSF.

Patients will undergo their ablative chemotherapy before transplantation. Patients will then be transplanted. The success of the transplantation will be evaluated. Graft durability will be evaluated to 12 months post-transplant. In the event that a sufficient number of cells for transplantation are not obtained from the collections, cells may be retained, pooled, and transplanted at a later date at the Investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to undergo autologous transplantation.
* Diagnosis of NHL, HD or MM [patients with plasma cell leukemia or other leukemias including chronic lymphocytic leukemia (CLL), are excluded].
* In the last collection attempt prior to entry into this trial, the patient has failed to collect 0.8x10^6 cells/kg in at least 2 apheresis sessions or 2x10^6 cells/kg in 4 apheresis sessions using a mobilization regimen of chemotherapy, with or without G-CSF.
* A minimum of a 7 day interval between last collection attempt and randomization.
* Cardiac, pulmonary and renal function deemed clinically adequate to be able to undergo mobilization and transplant.
* Performance status, Eastern Cooperative Oncology Group (ECOG) of 0 or 1
* ≥ 21 days between the last cycle of chemotherapy and randomization (thalidomide, dexamethasone, and other corticosteroids, Rituxan® and Velcade® are not considered prior chemotherapy for the purpose of this study).
* The patient has recovered from all acute toxic effects of prior chemotherapy.
* WBC ≥ 2.5x10^9/l.
* Absolute neutrophil count ≥ 1.5x10^9/l.
* Platelet count ≥ 75x10^9/l.
* Adequate renal function as demonstrated by serum creatine ≤ or equal to 2.2 mg/dl or creatinine clearance (24 hr urine collection)≥ 60 ml/min
* Serum Glutamate Oxaloacetate Transaminase (SGOT), Serum Glutamate Pyruvate Transaminase (SGPT) and total bilirubin ≤ 2.5 x upper limit of normal (ULN).
* Signed informed consent.
* All patients must agree to use a highly effective method of contraception (including both female patients of child-bearing potential and male patients with child-bearing potential partners). Effective birth control includes: a) birth control pills, depo-progesterone, or an IUD PLUS one barrier method, or b) two barrier methods. Effective barrier methods are: male and female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm). For patients using hormonal contraceptive method, information about any interaction of MAD3100 with hormonal contraceptives is not known.

Exclusion Criteria:

* A co-morbid condition which, in the view of the Investigators, renders the patient at high risk from treatment complications.
* A residual acute medical condition resulting from prior chemotherapy.
* Received thalidomide, dexamethasone or corticosteroids, Rituxan® and Velcade® within 7 days prior to randomization.
* Brain metastases or carcinomatous meningitis.
* Active acute or chronic infection or anti-infective therapy within 1 week prior to randomization.
* Fever (temperature ≥ 38 degrees celsius).
* Hypercalcemia (≥ 1mg/dl above the ULN).
* Known to be HIV-positive.
* Pregnant and nursing females.
* Patient unwilling to implement adequate birth control (including both female patients of child-bearing potential and male patients with child-bearing potential partners).
* Patients who previously received experimental therapy within 4 weeks of randomization or who are currently enrolled in another experimental protocol during the Mobilization phase.
* Patients who have failed previous collection attempt within 7 days or less from randomization.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-11; Primary Completion 2008-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To determine if patients reach a target of ≥ 2x10^6 CD34+ cells/kg within 2 days of apheresis in Non-Hodgkin's Lymphoma (NHL), Hodgkin's Disease (HD) or Multiple Myeloma (MM) patients who are proven poor mobilizer. | after last apheresis

SECONDARY OUTCOMES:
To examine and compare the safety of both mobilization regimens, G-CSF plus AMD3100(240µg/kg) and G-CSF plus placebo in NHL, MM and HD patients. | After each dose of AMD3100
To measure the daily and total number of CD34+ cells harvested during apheresis. | After each dose of AMD3100
To measure the number of days of apheresis needed to harvest ≥ 2x10^6 CD34+ cells/kg. | After each dose of AMD3100 transplantation and engraftment
To measure the number of days of apheresis needed to harvest ≥ 5x10^6 CD34+ cells/kg. | After each dose of AMD3100, transplantation and engraftment
To determine the times of platelet (PLT) and polymorphonuclear leukocyte (PMN) engraftment. | After each dose of AMD3100, transplantation and engraftment
To evaluate the durability of engraftment. | After each dose of AMD3100, transplantation and engraftment
To determine if patient reach the Optimum Target of 5x10^6 CD34+ cells/kg within 4 days of apheresis. | After each dose of AMD3100, transplantation and engraftment
To determine if NHL tumor cells are mobilized after either G-CSF mobilization of AMD3100 administration | After G-CSF mobilization period and after each dose of AMD3100

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (5):
- Germany (5):
  - Berlin
  - Cologne
  - Dresden
  - Nuremberg
  - Würzburg